CLINICAL TRIAL: NCT01528943
Title: The Effect of Prostacyclin on Haemostasis as Evaluated by Thrombelastography and Endothelial Markers in Patients Undergoing Major Abdominal Surgery. A Pilot Study
Brief Title: Effect of Prostacyclin on Haemostasis in Abdominal Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pär Johansson, Medical Director, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ET Abdominal
Record Dates: First submitted 2012-02-05; First posted 2012-02-08 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Surgery
Keywords: prostacycline, endothel integrity and abdominal surgery
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prostacyclin (Experimental): Treatment with prostacyclin
  Interventions: Drug: Prostacycline
- Isotonic saline (Placebo Comparator): Treatment with isotonic saline
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Prostacycline — Continuous infusion peri -and 6 hours postoperatively of prostacycline 1 ng/kg/min
  Arms: Prostacyclin
Drug: Isotonic saline — same volume as the group that are allocated to prostacycline
  Arms: Isotonic saline

SUMMARY:
The purpose of this study is to investigate the effect of continuous perioperative infusion of prostacyclin on haemostasis and endothelial functionality in patients undergoing major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women above 18 years old
* Undergoing Whipple surgery or liver resection
* Able and willing to give informed consent

Exclusion Criteria:

1. Allergy towards the study medication
2. In treatment with platelet ADP receptor inhibitors or heparin (not including thrombosis prophylaxis), Factor Xa inhibitors, trombininhibitors, Vitamin K antagonists
3. Autoimmune disease
4. Intracranial bleeding within the last 6 months
5. Acute coronary syndrome or myocardial infarction within the last 6 months
6. Congestive heart disease
7. Pregnant or breastfeeding
8. Participating in another clinical study within the last 30 days
9. Liver cirrhosis
10. Need for renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in endothelial biomarkers | Baseline to 6 hours postoperatively

SECONDARY OUTCOMES:
Functional haemostasis evaluated by thrombelastography | Baseline to 6 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Pär Johansson I Johansson, MD DMSc MPA, Principal Investigator — Professor
Locations (1):
- Rigshospitalet, Copenhagen, Region Sjælland, Denmark